CLINICAL TRIAL: NCT03843216
Title: End-growth Results of Tailored Treatment in 1938 Adolescents With High Risk Idiopathic Scoliosis: a Cohort Study From a Prospective Clinical Database
Brief Title: End Growth Results for Conservative Treatment for Idiopahitc Scoliosis
Status: Completed | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: EGR-ISICO
Record Dates: First submitted 2018-09-25; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Scoliosis; Adolescence; Scoliosis Idiopathic
MeSH Terms: conditions — Scoliosis | interventions — Observation; Braces

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — patients not treated
Other: Physiotherapic scoliosis specific exercise — Specific exercise according to the SEAS (Scientific Exercises Approach to Scoliosis) protocol
Device: brace — different kind of braces being elastic, rigid or very rigid. All devices are custom made. The hours of application per day varied from 18 to 24h.

SUMMARY:
This study evaluates in a prospectively collected multicenter cohort the existence, characteristics and determinants of EBPCA, the obtained results and their determinant, the rate of over- and under-treatment and their determinants.

DETAILED DESCRIPTION:
Since an evidence-based personalised conservative approach (EBPCA) to Adolescent Idiopathic Scoliosis has never been checked, the investigators studied a prospectively collected multicenter cohort with the aim to verify in the different clinical situations 1) the existence, characteristics and determinants of EBPCA; 2) the obtained results and their determinant; 3) the rate of over- and under-treatment and their determinants. These results are expected to check the actual evidence in everyday clinic, to provide a benchmark for future studies, and to inform guidelines producers and consequently health policy in high income countries, but also and particularly in low-middle income countries where surgery is difficult due to the high costs, and missing competences and structures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Adolescent Idiopathic Scoliosis (AIS),
* curves between 11 and 45° at start,
* Risser test between 0 and 2.
* Since our Institute receive many participants for a second opinion, we considered only participants in charge, defined as those who came at least three times to our facilities

Exclusion Criteria:

* previous bracing;
* absence of x-rays in the 3 months before/after the start and the end of treatment/observation.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Scoliotic patients that were referred to a tertiary clinic specialized on spine deformity.
Sampling Method: Non-Probability Sample
Enrollment: 1938 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving specific results | End of growth as defined as radiological evidence of Risser 5 or Risser 4 and two years of no growth in height.
  Outcomes were calculated as number of patients achieving specific results at the end of growth, including: 1) remaining below the significant prognostic thresholds of 30° and 50°; 2) improved or progressed beyond the measurement error of 5°; 3) achieving the treatment aims proposed by the current Guidelines : primary (optimal) and secondary (minimal); 4) receiving under- or over-treatment, that have been defined during study planning in relationship to the ideal final result.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Negrini, MD, Prof, Principal Investigator — stefano.negrini@isico.it
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17;369(16):1512-21. doi: 10.1056/NEJMoa1307337. Epub 2013 Sep 19. PMID 24047455
- [Background] Di Felice F, Zaina F, Donzelli S, Negrini S. The Natural History of Idiopathic Scoliosis During Growth: A Meta-Analysis. Am J Phys Med Rehabil. 2018 May;97(5):346-356. doi: 10.1097/PHM.0000000000000861. PMID 29493563
- [Background] Negrini S, Hresko TM, O'Brien JP, Price N; SOSORT Boards; SRS Non-Operative Committee. Recommendations for research studies on treatment of idiopathic scoliosis: Consensus 2014 between SOSORT and SRS non-operative management committee. Scoliosis. 2015 Mar 7;10:8. doi: 10.1186/s13013-014-0025-4. eCollection 2015. PMID 25780381